CLINICAL TRIAL: NCT01438593
Title: An Exploratory Clinical Trial to Assess Treatment of Chronic Ischemic Stroke With Brain Transplants of Purified CD34+ Umbilical Cord Blood Stem Cells
Brief Title: Study of Purified Umbilical Cord Blood CD34+ Stem Cell on Chronic Ischemic Stroke
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shinn-Zong Lin, Professor of Neurosurgery, China Medical University, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMR97-IRB-178-4
Record Dates: First submitted 2011-09-07; First posted 2011-09-22 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2011-12

CONDITIONS: Ischemic Stroke; Ischaemic Cerebral Infarction; Infarction, Middle Cerebral Artery; Ischemia; Brain Ischemia
Keywords: Stroke; Brain disease; Ischemia; Cerebral infraction; Cord Blood
MeSH Terms: conditions — Ischemic Stroke; Infarction, Middle Cerebral Artery; Ischemia; Brain Ischemia; Stroke; Brain Diseases | interventions — Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HUCB, Medicine, Rehabilitation (Experimental): Stroke patients are received intracerebral implantation of human cord blood stem cells (CD34+), Antiplatelet Medication, and Rehabilitation.
  Interventions: Procedure: Intercerebral implantation of allogenic CD34+ stem cell

INTERVENTIONS:
Procedure: Intercerebral implantation of allogenic CD34+ stem cell — Each patient will receive brain implant of approximately 5 million allogenic Umbilical cord blood CD34+ Stem Cell
  Other Names: Hematopoietic stem cell; Cord Blood Stem Cell; UCB Stem Cell

SUMMARY:
The purpose of the study is to determine the safety and possible effectiveness of brain transplants of CD34+ stem cells obtained from umbilical cord blood (UCB) to treat stroke.

DETAILED DESCRIPTION:
The study will use CD34+ cells (a special kind of cell that is believed to be a stem cell) isolated from UCB (blood obtained at birth from the umbilical cord blood of babies). StemCyte, a leading accredited UCB banking company with branches in the United States and Taiwan, will provide the units of UCB that match at least 5 out of 6 HLA (human leukocyte antigens) for transplantation. The HLA-matching is the same as that used to match cells and organs for transplantation so that the body does not reject the cells. We will isolate CD34 cells from these units, purified them, suspend the cells in solution (1 ml containing 2-8 million cells), and inject the cells into brain around the site damaged by the stroke

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can be of either gender and must be between 35 through 75 years of age.
2. Subjects must have had ischemic stroke more than 6 and less than 60 months ago.
3. Subjects must have stable hemiplegia or hemiparesis condition at least for 3 months.
4. Subjects must have stroke-induced clinical deficits affecting motor, perceptual, or language functions, with a National Institutes of Health Stroke Scale (NIHSS) of 5-15.
5. Subjects must have stroke in the middle cerebral artery territory.
6. Subjects must have an available umbilical cord blood unit that has an HLA-match of at least 5:6 (HLA-A, -B, and -DR).
7. Subjects must be able to read and understand the informed consent form that has been approved by the appropriate Institutional Review Board (IRB). The subject must sign and date the informed consent form before any study-specific procedures. (Note: If a subject consents to participation but is not in a position to sign and date the informed consent form personally because of his or her physical conditions, the consent form must be confirmed orally at the time of consent, marked or finger printed by the subject voluntarily). The informed consent procedure must be observed by an independent witness who is present throughout the whole informed consent process and sign the consent form.

Exclusion Criteria:

1. Subject has evidence of a non-ischemic mechanism, subarachnoid hemorrhage, primary intracerebral or intraventricular hemorrhage or MRI has shown that the occlusion is not in the middle cerebral artery territory.
2. Pregnant or lactating women.
3. History of alcohol or drug abuse in the previous 3 months.
4. Subjects must not have the following conditions in documents:

   * significant renal, cardiovascular, hepatic, or psychiatric disease
   * abnormal blood coagulation parameters,
   * immunodeficiency (e.g. AIDS)
   * tumors, leukemia, and other cancer that may interfere with the clinical trial protocol
   * infectious diseases, including hepatitis, or other conditions that may be a contraindication to the planned therapies and evaluation.
5. Subject must not be currently participating in another investigational study or taking any investigational drug within the last four weeks before the screening of this study.
6. Any other condition that, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol and would not be suitable to perform a surgery or to participate in the study.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in NIH Stroke Scale (NIHSS) | Change from baseline in NIHSS at 1 weeks
  Evaluate change from Baseline in NIHSS at 1 week
Change from Baseline in NIH Stroke Scale(NIHSS) | Change from Baseline in NIHSS at 2 weeks
  Evaluate change from Baseline in NIHSS at 2 weeks
Change from baseline in NIH Stroke Scale | Change from baseline in NIHSS at 4 weeks
  Evaluate change from baseline in NIHSS at 4 weeks
Change from baseline in NIH Stroke Scale ( NIHSS) | Change from baseline in NIHSS at 12 weeks
  Evaluate change from baseline in NIHSS at 12 weeks

SECONDARY OUTCOMES:
Change from baseline in Brain Image | Change from baseline in Brain Image at 1 week
  Brain Image will be performed by MRI. The MRI evaluation includes DEI, T1W, T2W, MRS, and DTI, and change from baseline will be evaluated at 1 week
Change from baseline in Brain Image | Change from baseline in Brain Image at 4 weeks
  Brain Image will be performed by MRI. The MRI evaluation includes DEI,T1W,T2W,MRS and DTI , and evaluate the change from baseline at 4 weeks
Change from baseline in Brain Image | Change from baseline in Brain Image at 6 months
  Brain Image will be performed by MRI.MRI image includes DEI,T1W, T2W, and DTI, and change from baseline will be evaluated at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shinn-Zong Lin, M.D.;PhD., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan, Taiwan